CLINICAL TRIAL: NCT06330103
Title: Assessing the Efficacy of Artificial Intelligence in Left Ventricular Function Screening Using Parasternal Long Axis View Cardiac Ultrasound Video Clips
Brief Title: Efficacy of AI EF Screening by Using Smartphone Application Recorded PLAX View Cardiac Ultrasound Video Clips
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rayong Hospital (Other)
Collaborators: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Sittiluck Wongwantanee, Principal Investigator, Rayong Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: RayongH
Record Dates: First submitted 2024-03-05; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Heart Failure; Heart Failure With Reduced Ejection Fraction; Cardiac Failure; Echocardiography; Artificial Intelligence
MeSH Terms: conditions — Heart Failure | interventions — Artificial Intelligence

STUDY DESIGN:
Intervention Model Description: 923 samples that were evaluated for LVEF by certified cardiologists, 739 clips were used to train AI, while the remaining 184 clips were used to test if AI could process the results correctly. Artificial intelligence aims to classify cardiac function into three groups: Reduced EF, Mildly Reduced EF, and Preserved LV.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LV function from cardiologist (Active Comparator): Certified Cardiologist will access and interpreted LV function by used traditional Echocardiography then separate result into three group Preserved LV ejection fraction(EF>50%), mildly reduce ejection fraction(EF40-49%), reduced LV ejection fraction(EF<40%)
  Interventions: Other: Easy EF
- LV function By artificial intelligence (Experimental): AI will access VDO clips in only parasternal long axis view and separate into three group Preserved LV ejection fraction(EF>50%), mildly reduce ejection fraction(EF40-49%), reduced LV ejection fraction(EF<40%)
  Interventions: Other: Easy EF

INTERVENTIONS:
Other: Easy EF — AI was integrated into the application smartphone and used smartphone camera to recorded shot VDO clip of heart ultrasound in parasternal long axis view and returned cardiac function result to user.
  Other Names: artificial intelligence; mobile smart phone application

SUMMARY:
Assessing the Efficacy of Artificial Intelligence in Left Ventricular Function Screening Using Parasternal Long Axis View Cardiac Ultrasound Video Clips

ABSTRACT BACKGROUND: Echocardiography serves as a fundamental diagnostic procedure for managing heart failure patients. Data from Thailand's Ministry of Public Health reveals that there is a substantial patient population, with over 100,000 admissions annually due to this condition. Nevertheless, the widespread implementation of echocardiography in this patient group remains challenging, primarily due to limitations in specialist resources, particularly in rural community hospitals. Although modern community hospitals are equipped with ultrasound machines capable of basic cardiac assessment (e.g., parasternal long axis view), the demand for expert cardiologists remains a formidable obstacle to achieving comprehensive diagnostic capabilities. Leveraging the capabilities of Artificial Intelligence (AI) technology, proficient in the accurate prediction and processing of diverse healthcare data types, offers a promising for addressing this prevailing issue. This study is designed to assess the effectiveness of AI in evaluating cardiac performance from parasternal long axis view ultrasound video clips obtained via the smartphone application.

OBJECTIVES: To evaluate the effectiveness of artificial intelligence in screening cardiac function from parasternal long axis view cardiac ultrasound video clips obtained through the smartphone application.

DETAILED DESCRIPTION:
METHODS: The investigators built the smartphone application to collect parasternal long axis view video clips and used artificial intelligence "Easy EF" to evaluate cardiac function. All samples that were evaluated for LVEF by certified cardiologists, 70% of all clips were used to train AI, while the remaining 30% of clips were used to test if AI could process the results correctly. Artificial intelligence aims to classify cardiac function into three groups: Reduced EF, Mildly Reduced EF, and Preserved LV.

ELIGIBILITY:
Inclusion Criteria:

* Shot 5 second VDO clip of Parasternal long axis heart ultrasound recorded by smartphone Application "Easy EF" without patient identification with result of Ejection fraction that performed by certify cardiologist approved result

Exclusion Criteria:

* Incomplete VDO clip (too much shaking, too shot recording)
* Lighting was inappropriate
* Inappropriate ultrasound framing
* arrhythmia (atrial fibrillation)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 923 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
efficiency of AI in screening left ventricular cardiac function by use smartphone application | 3 month
  percentage of correct LV function clip that interpreted by AI in each LV function group(Preserved LV, Mildly reduced LV, Reduced LV function) and overall compare with result from certified cardiologist

CONTACTS AND LOCATIONS:
Locations (1):
- Rayong Hospital, Rayong, Thailand

IPD SHARING:
Plan to Share IPD: Yes
result of AI screening
Supporting Information: Study Protocol, SAP
Time Frame: 3 month
Access Criteria: contact rayong hospital